CLINICAL TRIAL: NCT04658186
Title: A Double-Blind, Placebo-Controlled, Randomized, 18-Month Phase 2a Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Oral UCB0599 in Study Participants With Early Parkinson's Disease
Brief Title: A 18-month Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Oral UCB0599 in Study Participants With Early-stage Parkinson's Disease
Acronym: ORCHESTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Collaborators: The Parkinson Study Group (Network)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PD0053; 2020-003265-19 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Early-stage Parkinson's Disease
Keywords: Early-stage parkinson's disease; UCB0599; Phase 2; Early-stage PD
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- UCB0599 High Dose Arm (Experimental): Participants will be randomized to receive a predefined high dosage of UCB0599 during the Treatment Period.
  Interventions: Drug: UCB0599
- Placebo Arm (Placebo Comparator): Participants will be randomized to receive a predefined dosage of Placebo during the Treatment Period.
  Interventions: Drug: Placebo
- UCB0599 Low Dose Arm (Experimental): Participants will be randomized to receive a predefined low dosage of UCB0599 during the Treatment Period.
  Interventions: Drug: UCB0599

INTERVENTIONS:
Drug: UCB0599 — Drug: UCB0599 Pharmaceutical form: Granules in capsules Route of administration: Oral use Participants will receive UCB0599 in a pre-specified sequence during the Treatment Period.
  Arms: UCB0599 High Dose Arm; UCB0599 Low Dose Arm
Drug: Placebo — Drug: Placebo Pharmaceutical form: Capsules Route of administration: Oral use Participants will receive Placebo in a pre-specified sequence during the Treatment Period.
  Arms: Placebo Arm

SUMMARY:
The purpose of the study is to assess the safety and tolerability of UCB0599 and to demonstrate the superiority of UCB0599 over placebo with regard to clinical symptoms of disease progression over 12 and 18 months in participants diagnosed with early-stage Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be 40 to 75 years of age inclusive, at the time of signing the informed consent
* Study participant has Parkinson's Disease (PD), with a diagnosis made by a neurologist according to the 2015 Movement Disorder Society criteria within 2 years of Baseline Visit (including diagnosis during Screening)
* The following diagnostic criteria must be met: bradykinesia AND at least ONE of the following: muscular rigidity, or resting tremor
* A Screening Dopamine Transporter Imaging with Single Photon Emission Computed Tomography (DaT-SPECT), or a historical DaT-SPECT within 3 months of the Screening Visit that has been qualified by the central reader, shows evidence of dopamine transporter deficit per study requirements and as determined by a central reader
* Study participant is in the ≤2.5 modified Hoehn and Yahr stage at Screening
* Study participant has never taken medications for the treatment of motor symptoms of PD and is not expected to require starting symptomatic treatment (ST) with a high likelihood in the next 6 months as far as clinical judgement allows
* Study participant has never taken part in disease-modifying treatment studies directed at neurodegenerative disease (NDD)
* Study participant does not take N-acetyl cysteine or other cysteine donors or glutathione precursors on a regular basis as a food supplement
* Study participant is willing, competent, and able to comply with all aspects of the protocol, including follow-up schedule and biospecimen collection
* Study participant has a body mass index (BMI) of 16 to 34kg/m² (inclusive)
* Contraception i) A male participant must agree to use contraception during the Treatment Period and for at least 90 days after the last dose ofstudy medication and refrain from donating sperm during this period ii) A female participant is eligible to participate if she is not pregnant, not breastfeeding, andat least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the Treatment Period and for at least 1 month after the last dose of study medication. The study participant must have a negative serum pregnancy test at Screening, which is to be confirmed negative by urine testing prior to the first dose of study medication at Baseline (Visit 3). If oral contraception is used, an additional barrier method will be required during the study as a study medication related-gastrointestinal upset or a drug interaction by CYP3A4 induction could interfere with efficacy

Exclusion Criteria:

* Study participant has a known hypersensitivity to any components (and/or its excipients) of the study medication or comparative drugs as stated in the protocol
* Study participant has a brain magnetic resonance imaging (MRI) scan performed during Screening indicative of a clinically significant abnormality or a historical MRI scan during the 6 months before Screening Visit 1 of sufficient quality to show such abnormalities. In case of doubt, the significance is determined on a case-by-case basis in close collaboration with the Medical Monitor and should not include abnormalities like age-appropriate brain atrophy, minor white matter signals, or mild vasculopathy
* Study participant has any contraindication for the brain MRI or Dopamine Transporter Imaging with Single Photon Emission Computed Tomography (DaT-SPECT) imaging
* Study participant has a Montreal Cognitive Assessment (MoCA) score less than 23, indicating mild cognitive impairment or other significant cognitive impairment or clinical dementia at Screening that, in the opinion of the Investigator, would interfere with study evaluation
* Study participant has abnormalities in lumbar spine previously known or determined by a Screening lumbar x-ray (if conducted) that could preclude lumbar puncture, in the opinion of the Investigator. The participant must be excluded from lumbar puncture but not from study participation
* Study participant has clinically significant electrocardiogram (ECG) abnormality at Screening, in the opinion of the Investigator
* Study participant has past history of use of medications for the treatment of motor symptoms of PD. Short (up to 4 weeks) past use of medications for the treatment of motor symptoms is permitted following a sufficient washout period. Medications included are: levodopa (maximum 400mg per day), dopamine agonists, monoamine oxidase B (MAO-B) inhibitors, anticholinergics, or amantadine. A sufficient washout period is at least 3 months prior to the Baseline Visit

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (115):
- United States (57):
  - Pd0053 50140, Birmingham, Alabama
  - Pd0053 50506, Phoenix, Arizona
  - Pd0053 50081, Phoenix, Arizona
  - Pd0053 50391, Tucson, Arizona
  - Pd0053 50539, Little Rock, Arkansas
  - Pd0053 50519, Fountain Valley, California
  - Pd0053 50385, Fresno, California
  - Pd0053 50416, La Jolla, California
  - Pd0053 50118, Los Angeles, California
  - Pd0053 50531, Englewood, Colorado
  - Pd0053 50392, Danbury, Connecticut
  - Pd0053 50538, Farmington, Connecticut
  - Pd0053 50396, Boca Raton, Florida
  - Pd0053 50524, Bradenton, Florida
  - Pd0053 50199, Miami, Florida
  - Pd0053 50394, Tampa, Florida
  - Pd0053 50544, Augusta, Georgia
  - Pd0053 50401, Chicago, Illinois
  - Pd0053 50310, Chicago, Illinois
  - Pd0053 50399, Winfield, Illinois
  - Pd0053 50549, Iowa City, Iowa
  - Pd0053 50074, Kansas City, Kansas
  - Pd0053 50121, Lexington, Kentucky
  - Pd0053 50395, New Orleans, Louisiana
  - Pd0053 50529, Baltimore, Maryland
  - Pd0053 50547, Baltimore, Maryland
  - Pd0053 50243, Boston, Massachusetts
  - Pd0053 50546, Worcester, Massachusetts
  - Pd0053 50386, Farmington Hills, Michigan
  - Pd0053 50536, Saint Paul, Minnesota
  - Pd0053 50397, Las Vegas, Nevada
  - Pd0053 50299, New Brunswick, New Jersey
  - Pd0053 50077, New York, New York
  - Pd0053 50521, New York, New York
  - Pd0053 50119, New York, New York
  - Pd0053 50530, Stony Brook, New York
  - Pd0053 50535, Williamsville, New York
  - Pd0053 50372, Cleveland, Ohio
  - Pd0053 50311, Cleveland, Ohio
  - Pd0053 50255, Columbus, Ohio
  - Pd0053 50527, Toledo, Ohio
  - Pd0053 50398, Tulsa, Oklahoma
  - Pd0053 50510, Portland, Oregon
  - Pd0053 50526, Philadelphia, Pennsylvania
  - Pd0053 50084, Charleston, South Carolina
  - Pd0053 50532, Knoxville, Tennessee
  - Pd0053 50543, Memphis, Tennessee
  - Pd0053 50525, Houston, Texas
  - Pd0053 50113, Houston, Texas
  - Pd0053 50400, San Antonio, Texas
  - Pd0053 50107, Burlington, Vermont
  - Pd0053 50542, Charlottesville, Virginia
  - Pd0053 50410, Fairfax, Virginia
  - Pd0053 50534, Virginia Beach, Virginia
  - Pd0053 50292, Kirkland, Washington
  - Pd0053 50419, Spokane, Washington
  - Pd0053 50402, Crab Orchard, West Virginia
- Canada (4):
  - Pd0053 50374, Calgary
  - Pd0053 50390, Kelowna
  - Pd0053 50387, Ottawa
  - Pd0053 50389, Toronto
- France (10):
  - Pd0053 40197, Amiens
  - Pd0053 40527, Bordeaux
  - Pd0053 40424, Créteil
  - Pd0053 40526, Lille
  - Pd0053 40130, Marseille
  - Pd0053 40635, Nantes
  - Pd0053 40524, Nîmes
  - Pd0053 40525, Paris
  - Pd0053 40131, Strasbourg
  - Pd0053 40528, Toulouse
- Germany (12):
  - Pd0053 40515, Berlin
  - Pd0053 40138, Bonn
  - Pd0053 40530, Dresden
  - Pd0053 40711, Erbach im Odenwald
  - Pd0053 40023, Erlangen
  - Pd0053 40710, Essen
  - Pd0053 40532, Haag in Oberbayern
  - Pd0053 40024, Hanover
  - Pd0053 40249, Kiel
  - Pd0053 40174, Mainz
  - Pd0053 40529, Marburg
  - Pd0053 40531, Regensburg
- Italy (5):
  - Pd0053 40555, Brescia
  - Pd0053 40533, Padua
  - Pd0053 40257, Roma
  - Pd0053 40534, Roma
  - Pd0053 40697, Roma
- Pd0053 40359, Nijmegen, Netherlands
- Poland (11):
  - Pd0053 40694, Bydgoszcz
  - Pd0053 40719, Jelenia Góra
  - Pd0053 40539, Katowice
  - Pd0053 40538, Krakow
  - Pd0053 40696, Krakow
  - Pd0053 40700, Lodz
  - Pd0053 40702, Lublin
  - Pd0053 40535, Oświęcim
  - Pd0053 40536, Warsaw
  - Pd0053 40699, Warsaw
  - Pd0053 40705, Warsaw
- Spain (9):
  - Pd0053 40045, A Coruña
  - Pd0053 40159, Barcelona
  - Pd0053 40267, Barcelona
  - Pd0053 40046, Córdoba
  - Pd0053 40540, Madrid
  - Pd0053 40542, Móstoles
  - Pd0053 40352, Pamplona
  - Pd0053 40541, San Sebastián
  - Pd0053 40049, Seville
- United Kingdom (6):
  - Pd0053 40175, London
  - Pd0053 40543, London
  - Pd0053 40698, London
  - Pd0053 40544, Motherwell
  - Pd0053 40306, Newcastle upon Tyne
  - Pd0053 40457, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/

REFERENCES:
- [Derived] Price DL, Khan A, Angers R, Cardenas A, Prato MK, Bani M, Bonhaus DW, Citron M, Biere AL. In vivo effects of the alpha-synuclein misfolding inhibitor minzasolmin supports clinical development in Parkinson's disease. NPJ Parkinsons Dis. 2023 Jul 17;9(1):114. doi: 10.1038/s41531-023-00552-7. PMID 37460603

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in December 2020 and concluded in September 2024.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants received UCB0599 matching-placebo capsules, orally, from Day 1 up to 18 months during treatment period.
- UCB0599 180 mg/Day: Participants received UCB0599 90 milligram (mg) capsules twice daily (BID), for a total daily dose of 180 mg, along with matching placebo capsules BID, administered orally from Day 1 up to 18 months during treatment period.
- UCB0599 360 mg/Day: Participants received UCB0599 180 mg capsules twice daily (BID), for a total daily dose of 360 mg, administered orally from Day 1 up to 18 months during treatment period.
Period: Overall Study
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Started | 165 | 166 | 165
Completed | 154 | 138 | 139
Not Completed | 11 | 28 | 26
Not completed — Adverse Event | 4 | 18 | 15
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Participant Not Eligible. Randomized In Error | 1 | 0 | 1
Not completed — Participant is Moving in Another Province | 0 | 1 | 0
Not completed — Non-Compliance | 0 | 1 | 1
Not completed — Site Closure; Participant declined transfer | 0 | 1 | 0
Not completed — Dropout on the Promotor's Decision | 0 | 0 | 1
Not completed — Worsening Symptoms; Participant Withdrew | 0 | 0 | 1
Not completed — PI Decision due to Participant Safety | 0 | 0 | 1
Not completed — Consent Withdrawn by Participant (not due to adverse event) | 5 | 6 | 3

BASELINE CHARACTERISTICS:
Population: The randomized set (RS) included all study participants who are randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day | Total
Number analyzed (Participants) | 165 | 166 | 165 | 496
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.3) | 61.4 (7.8) | 59.9 (8.4) | 60.8 (8.2)
Age, Customized [Count of Participants; unit: Participants]
  18 years to less than (<) 65 years | 98 | 105 | 110 | 313
  65 years to <85 years | 67 | 61 | 55 | 183
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 66 | 65 | 196
  Male | 100 | 100 | 100 | 300
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 1 | 1 | 4
  Race: White | 134 | 143 | 143 | 420
  Race: Other/Mixed | 4 | 0 | 2 | 6
  Race: Missing | 25 | 22 | 19 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 4 | 3 | 5 | 12
  Ethnicity: Not Hispanic or Latino | 136 | 141 | 141 | 418
  Ethnicity: Missing | 25 | 22 | 19 | 66

OUTCOME MEASURES:

1. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Day 0
Description: MDS-UPDRS is a multimodal scale. Part I assessed non-motor experiences of daily living and has 2 components (0-52 possible points). Part IA contains 6 questions and is assessed by the examiner (0-24 possible points). Part IB contains 7 questions on non-motor experiences of daily living completed by participant (0-28 possible points). Part II assessed motor experiences of daily living (0-52 possible points) and includes 13 questions completed by participant. Part III assessed motor signs of PD and was administered by rater (0-52 possible points). Part III contained 33 questions based on 18 items. For all questions of each part, numeric score response options linked to accepted clinical terms: 0 to 4, 0=Normal, 1=Slight, 2=Mild, 3=Moderate, 4=Severe. Total Score equals sum of Parts I, II, and III (Score: 0-236). Higher score = more severe PD symptoms.
Time Frame: Day 0
Population: Full analysis set (FAS) included all randomized study participants who received at least a partial dose of study medication, have at least 1 post-Baseline assessment. Here, number of participants analyzed included all participants who were evaluable for this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 156 | 159 | 159
score on a scale | 34.0 (13.2) | 33.9 (16.4) | 30.6 (13.4)

2. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 2
Description: as for outcome 1
Time Frame: Month 2
Population: FAS included all randomized study participants who received at least a partial dose of study medication, have at least 1 post-Baseline assessment. Here, number of participants analyzed included all participants who were evaluable for this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 153 | 156 | 144
score on a scale | 34.7 (13.9) | 34.8 (18.0) | 30.3 (14.6)

3. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 4
Description: as for outcome 1
Time Frame: Month 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 153 | 148 | 143
score on a scale | 34.7 (14.9) | 34.3 (18.6) | 31.4 (15.0)

4. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 6
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 154 | 147 | 146
score on a scale | 37.9 (16.0) | 36.6 (20.0) | 32.9 (15.7)

5. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 8
Description: as for outcome 1
Time Frame: Month 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 155 | 148 | 143
score on a scale | 35.6 (14.3) | 34.6 (19.7) | 32.9 (15.5)

6. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 10
Description: as for outcome 1
Time Frame: Month 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 156 | 141 | 140
score on a scale | 35.6 (13.6) | 33.7 (18.4) | 33.2 (15.6)

7. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 12
Description: as for outcome 1
Time Frame: Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 152 | 142 | 140
score on a scale | 37.3 (15.3) | 36.5 (19.2) | 34.5 (15.4)

8. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 14
Description: as for outcome 1
Time Frame: Month 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 154 | 137 | 141
score on a scale | 37.1 (14.6) | 34.8 (18.8) | 33.9 (16.9)

9. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 16
Description: as for outcome 1
Time Frame: Month 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 152 | 139 | 137
score on a scale | 37.2 (15.6) | 35.9 (19.8) | 33.6 (15.4)

10. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-III Sum Score at Month 18
Description: as for outcome 1
Time Frame: Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 152 | 138 | 137
score on a scale | 37.9 (15.5) | 35.6 (18.1) | 34.9 (16.4)

11. Secondary Outcome: MDS-UPDRS Part III Subscale
Description: MDS-UPDRS part III includes motor items assessing speech, facial expression, rigidity, finger tapping, hand movements, pronation supination movements of hands, toe tapping, leg agility, arising from chair, gait, freezing of gait, postural stability, posture, global spontaneity of movement (body bradykinesia), postural tremor of the hands, kinetic tremor of the hands, rest tremor amplitude, and constancy of rest tremor. It included 33 scores based on 18-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range was from 0 to 132, with a lower score indicating better motor function and a higher score indicating more severe motor symptoms.
Time Frame: Day 0, Months 2, 4, 6, 8, 10, 12, 14, 16, 18
Population: FAS included all randomized study participants who received at least a partial dose of study medication, have at least 1 post-Baseline assessment. Here, number of participants analyzed included all participants who were evaluable for this assessment and number analyzed (n) signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 159 | 162 | 164
score on a scale
  Day 0 | 22.6 (9.8) | 21.9 (11.3) | 20.4 (9.5)
  Month 2: number analyzed (Participants) | 159 | 158 | 151
  Month 2 | 22.9 (10.2) | 22.7 (12.4) | 20.0 (10.3)
  Month 4: number analyzed (Participants) | 157 | 151 | 147
  Month 4 | 23.1 (10.5) | 22.5 (12.7) | 20.7 (10.6)
  Month 6: number analyzed (Participants) | 157 | 147 | 147
  Month 6 | 24.3 (10.9) | 23.2 (12.4) | 21.3 (10.8)
  Month 8: number analyzed (Participants) | 156 | 148 | 145
  Month 8 | 23.3 (10.0) | 22.2 (12.6) | 21.0 (10.7)
  Month 10: number analyzed (Participants) | 156 | 141 | 140
  Month 10 | 23.3 (9.2) | 21.6 (12.1) | 21.0 (11.0)
  Month 12: number analyzed (Participants) | 153 | 143 | 140
  Month 12 | 24.1 (10.0) | 22.8 (12.0) | 21.8 (10.5)
  Month 14: number analyzed (Participants) | 154 | 139 | 141
  Month 14 | 24.1 (10.1) | 22.2 (11.9) | 21.8 (11.4)
  Month 16: number analyzed (Participants) | 153 | 139 | 137
  Month 16 | 24.3 (10.1) | 22.8 (12.3) | 21.7 (10.7)
  Month 18: number analyzed (Participants) | 153 | 138 | 138
  Month 18 | 24.2 (10.1) | 23.0 (11.7) | 22.2 (10.9)

12. Secondary Outcome: MDS-UPDRS Part III Early-stage Parkinson's Disease (ePD) Subscore on Selected Items
Description: The early-stage Parkinson's disease (ePD) subscore is derived from a 15-item subset of the MDS-UPDRS Part III (Motor Examination). It includes all rigidity assessments (neck, upper limbs [right/left], and lower limbs [right/left]) and bradykinesia-related tasks: finger tapping (right/left), hand movements (right/left), pronation-supination of hands (right/left), toe tapping (right/left), and leg agility (right/left). Each item is scored on a 5-point likert scale (0 = no problem to 4 = severe), resulting in a total ePD subscore range of 0 to 60. Higher scores indicate greater motor impairment, while lower scores reflect better motor function.
Time Frame: Day 0, Months 2, 4, 6, 8, 10, 12, 14, 16, 18
Population: FAS included all randomized study participants who received at least a partial dose of study medication, have at least 1 post-Baseline assessment. Here, number of participants analyzed included all participants who were evaluable for this assessment and 'n' signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 159 | 162 | 164
score on a scale
  Day 0 | 13.3 (7.11) | 12.6 (7.96) | 11.8 (6.85)
  Month 2: number analyzed (Participants) | 159 | 159 | 151
  Month 2 | 13.2 (7.33) | 13.2 (8.48) | 11.6 (7.57)
  Month 4: number analyzed (Participants) | 157 | 151 | 147
  Month 4 | 13.4 (7.50) | 13.1 (8.76) | 11.8 (7.64)
  Month 6: number analyzed (Participants) | 157 | 148 | 147
  Month 6 | 13.9 (7.39) | 13.4 (8.42) | 12.4 (7.58)
  Month 8: number analyzed (Participants) | 157 | 148 | 146
  Month 8 | 13.4 (6.82) | 12.7 (8.60) | 11.8 (7.49)
  Month 10: number analyzed (Participants) | 156 | 141 | 141
  Month 10 | 13.4 (6.46) | 12.1 (8.14) | 11.9 (7.98)
  Month 12: number analyzed (Participants) | 153 | 144 | 142
  Month 12 | 13.7 (6.98) | 12.7 (8.20) | 12.9 (7.61)
  Month 14: number analyzed (Participants) | 154 | 142 | 141
  Month 14 | 13.8 (7.14) | 12.7 (8.35) | 12.5 (7.88)
  Month 16: number analyzed (Participants) | 153 | 139 | 138
  Month 16 | 13.8 (7.24) | 12.9 (8.26) | 12.4 (7.83)
  Month 18: number analyzed (Participants) | 153 | 138 | 138
  Month 18 | 13.8 (7.34) | 12.9 (7.90) | 12.6 (7.61)

13. Secondary Outcome: MDS-UPDRS Part II Subscale
Description: MDS-UPDRS part II includes motor items assessing speech, saliva and drooling, chewing and swallowing, eating tasks (cutting food and handling utensils), dressing, hygiene, handwriting, doing hobbies and other activities, turning in bed, tremor, getting out of bed, a car or a deep chair, walking and balance, and freezing. Each of the items in the UPDRS is measured on a scale. It included 13-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range for Part II was 0-52, with higher scores reflecting greater severity.
Time Frame: Day 0, Months 2, 4, 6, 8, 10, 12, 14, 16, 18
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 163 | 163 | 161
score on a scale
  Day 0 | 6.0 (4.0) | 6.3 (4.6) | 5.7 (4.3)
  Month 2: number analyzed (Participants) | 158 | 160 | 149
  Month 2 | 6.5 (4.3) | 6.9 (5.2) | 6.1 (4.1)
  Month 4: number analyzed (Participants) | 156 | 150 | 147
  Month 4 | 6.8 (4.6) | 7.1 (5.4) | 6.4 (4.5)
  Month 6: number analyzed (Participants) | 156 | 148 | 147
  Month 6 | 7.7 (5.1) | 7.7 (6.2) | 6.7 (5.0)
  Month 8: number analyzed (Participants) | 158 | 148 | 145
  Month 8 | 7.0 (4.6) | 7.1 (5.7) | 6.9 (4.7)
  Month 10: number analyzed (Participants) | 156 | 142 | 143
  Month 10 | 6.9 (4.5) | 6.7 (5.4) | 7.1 (4.7)
  Month 12: number analyzed (Participants) | 153 | 144 | 143
  Month 12 | 6.9 (4.9) | 7.3 (5.5) | 7.3 (5.1)
  Month 14: number analyzed (Participants) | 154 | 140 | 142
  Month 14 | 7.1 (4.8) | 7.2 (5.8) | 7.0 (5.1)
  Month 16: number analyzed (Participants) | 152 | 140 | 138
  Month 16 | 7.1 (5.1) | 7.2 (5.7) | 6.7 (4.5)
  Month 18: number analyzed (Participants) | 152 | 138 | 138
  Month 18 | 7.3 (5.0) | 6.8 (5.2) | 7.3 (5.3)

14. Secondary Outcome: MDS-UPDRS Part I Subscale
Description: MDS-UPDRS part I include several non-motor aspects of experiences of daily living including cognitive impairment, hallucinations and psychosis, depressed mood, anxious mood, apathy, features of dopamine dysregulation syndrome during part 1A and sleep problems, daytime sleepiness, pain and other sensation, urinary problems, constipation problems, lightheadedness on standing, and fatigue during Part 1B. Part I assessed non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contained 6 questions and were assessed by examiner (Range 0-24). Part IB contained 7 questions on non-motor experiences of daily living which were completed by participant (Range 0-28). Each of items in UPDRS is measured on a scale of 0 to 4, where 0 is normal and 4 (higher score) represents severe abnormalities/worse outcome. Total Score Range 0 to 52. Total score is sum of Part IA (0-24) and Part IB (0-28) subscale scores. Higher scores indicated greater severity of non-motor symptoms.
Time Frame: Day 0, Months 2, 4, 6, 8, 10, 12, 14, 16, 18
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 158 | 161 | 158
score on a scale
  Day 0 | 5.4 (3.9) | 5.5 (4.4) | 4.7 (3.7)
  Month 2: number analyzed (Participants) | 155 | 160 | 145
  Month 2 | 5.2 (4.2) | 5.2 (3.8) | 4.3 (3.5)
  Month 4: number analyzed (Participants) | 153 | 149 | 144
  Month 4 | 5.1 (4.4) | 5.0 (4.0) | 4.5 (3.8)
  Month 6: number analyzed (Participants) | 154 | 148 | 146
  Month 6 | 5.9 (4.8) | 5.7 (4.5) | 5.1 (3.9)
  Month 8: number analyzed (Participants) | 156 | 148 | 147
  Month 8 | 5.5 (4.4) | 5.3 (4.2) | 5.0 (3.9)
  Month 10: number analyzed (Participants) | 156 | 142 | 143
  Month 10 | 5.4 (4.2) | 5.4 (4.1) | 4.9 (4.1)
  Month 12: number analyzed (Participants) | 152 | 143 | 143
  Month 12 | 6.2 (5.1) | 6.2 (4.8) | 5.3 (4.4)
  Month 14: number analyzed (Participants) | 154 | 141 | 142
  Month 14 | 5.9 (4.6) | 5.8 (5.0) | 5.0 (4.2)
  Month 16: number analyzed (Participants) | 153 | 140 | 138
  Month 16 | 5.9 (4.8) | 5.9 (5.1) | 5.1 (4.1)
  Month 18: number analyzed (Participants) | 152 | 138 | 138
  Month 18 | 6.4 (5.1) | 5.9 (4.6) | 5.3 (4.5)

15. Secondary Outcome: Emerging Symptoms in Participants as Measured by MDS-UPDRS Part II
Description: The participant was considered to have an emerging symptom for the item, if the change from Baseline for the item is greater than 0 for 2 consecutive visits. The magnitude of change from Baseline was not considered to determine the emerging symptom. Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part II includes motor items assessing speech, saliva and drooling, chewing and swallowing, eating tasks (cutting food and handling utensils), dressing, hygiene, handwriting, doing hobbies and other activities, turning in bed, tremor, getting out of bed, a car or a deep chair, walking and balance, and freezing. This included 13-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range for Part II was 0-52, with higher scores reflecting greater severity.
Time Frame: Baseline to Month 18
Population: FAS included all randomized study participants who received at least a partial dose of study medication, have at least 1 post-Baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 163 | 164 | 164
Participants
  Number of Emerging symptoms: 0 | 28 | 36 | 38
  Number of Emerging symptoms: 1 | 18 | 41 | 31
  Number of Emerging symptoms: 2 | 35 | 33 | 23
  Number of Emerging symptoms: 3 | 37 | 15 | 26
  Number of Emerging symptoms: 4 | 15 | 13 | 15
  Number of Emerging symptoms: 5 | 15 | 13 | 14
  Number of Emerging symptoms: 6 | 4 | 7 | 10
  Number of Emerging symptoms: 7 | 4 | 4 | 4
  Number of Emerging symptoms: 8 | 4 | 1 | 3
  Number of Emerging symptoms: 9 | 2 | 1 | 0
  Number of Emerging symptoms: 10 | 1 | 0 | 0
  Number of Emerging symptoms: 11 | 0 | 0 | 0
  Number of Emerging symptoms: 12 | 0 | 0 | 0
  Number of Emerging symptoms: 13 | 0 | 0 | 0

16. Secondary Outcome: Time to Worsening of the Disease as Measured by MDS-UPDRS Part III
Description: Time to worsening of the disease on the MDS-UPDRS III scale as defined by a 5-point increase in MDS-UPDRS III, within the 18-month period. MDS-UPDRS part III includes motor items assessing speech, facial expression, rigidity, finger tapping, hand movements, pronation supination movements of hands, toe tapping, leg agility, arising from chair, gait, freezing of gait, postural stability, posture, global spontaneity of movement (body bradykinesia), postural tremor of the hands, kinetic tremor of the hands, rest tremor amplitude, and constancy of rest tremor. It included 33 scores based on 18-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range was from 0 to 132, with a lower score indicating better motor function and a higher score indicating more severe motor symptoms.
Time Frame: Baseline to Month 18
Population: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 163 | 164 | 164
months | 8.64 [7.7236 to 9.5635] | 8.95 [7.8974 to 10.0012] | 9.45 [8.4743 to 10.4340]
Statistical Analysis 1: Comparison: Placebo vs UCB0599 180 mg/Day; Test type: Superiority; p = 0.647, Wald Chi-square; Difference in RMET = 0.31, 95% CI 2-sided [-1.00 to 1.61] — Results were obtained from a generalized linear model for the restricted mean event time (RMET), with gender and age at baseline as covariates and treatment group as the effect of interest
Statistical Analysis 2: Comparison: Placebo vs UCB0599 360 mg/Day; Test type: Superiority; p = 0.214, Wald Chi-square; Difference in RMET = 0.81, 95% CI 2-sided [-0.47 to 2.09] — Results obtained from generalized linear model for RMET, with gender and age at baseline as covariates and treatment group as effect of interest

17. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) is a standardized screening tool used to evaluate mild cognitive impairment across multiple cognitive functions i.e. visuospatial/executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. The total possible score is calculated by summing the scores across all functions ranges from: 0 to 30. A score of 26 or above is considered normal, a lower score indicates cognitive impairment.
Time Frame: Screening, Month 18
Population: FAS included all randomized study participants who received at least a partial dose of study medication, have at least 1 post-Baseline assessment. Here, 'n' signifies participants who were evaluable at each specified timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 163 | 164 | 164
score on a scale
  Screening | 27.8 (1.8) | 27.6 (2.0) | 27.8 (1.7)
  Month 18: number analyzed (Participants) | 152 | 137 | 136
  Month 18 | 27.4 (2.2) | 27.3 (2.4) | 27.3 (2.4)

18. Secondary Outcome: Change From Screening in Dopamine Transporter Imaging With Single Photon Emission Computed Tomography (DaT-SPECT) Mean Striatum Specific Binding Ratios (SBR)
Description: The change from screening in mean striatum specific binding ratios (SBR) was assessed by DaT-SPECT using 123I-Ioflupane as radiopharmaceutical. The whole striatum was calculated as the average of the SBR data values for the four following "small" regions: left caudate small, left putamen small, right caudate small and right putamen small. The SBR was calculated for each region with the occipital cortex as a reference region, where a lower SBR indicates worse disease. The following formula was used to calculate this: (Average [Small region] - Average [Occipital region])/ (Average [Occipital region]).
Time Frame: Screening, Months 12 and 18
Population: FAS included all randomized study participants who received at least a partial dose of study medication, have at least 1 post-Baseline assessment. Here, number of participants analyzed included all participants who were evaluable for this assessment and 'n' signifies participants who were evaluable at each specified timepoints.
Measure: Mean (Standard Deviation); unit: specific binding ratio
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 140 | 133 | 130
specific binding ratio
  Whole striatum: Month 12: number analyzed (Participants) | 133 | 130 | 111
  Whole striatum: Month 12 | -0.202 (0.215) | -0.141 (0.194) | -0.102 (0.254)
  Whole striatum: Month 18: number analyzed (Participants) | 140 | 124 | 130
  Whole striatum: Month 18 | -0.233 (0.226) | -0.182 (0.232) | -0.193 (0.254)
  Ipsilateral striatum: Month 12: number analyzed (Participants) | 114 | 114 | 95
  Ipsilateral striatum: Month 12 | -0.237 (0.262) | -0.161 (0.246) | -0.093 (0.294)
  Ipsilateral striatum: Month 18: number analyzed (Participants) | 123 | 109 | 114
  Ipsilateral striatum: Month 18 | -0.260 (0.263) | -0.211 (0.282) | -0.194 (0.318)
  Contralateral striatum: Month 12: number analyzed (Participants) | 114 | 114 | 95
  Contralateral striatum: Month 12 | -0.161 (0.210) | -0.138 (0.209) | -0.099 (0.278)
  Contralateral striatum: Month 18: number analyzed (Participants) | 123 | 109 | 114
  Contralateral striatum: Month 18 | -0.203 (0.214) | -0.169 (0.237) | -0.188 (0.259)
  Ipsilateral caudate small: Month 12: number analyzed (Participants) | 114 | 114 | 95
  Ipsilateral caudate small: Month 12 | -0.296 (0.380) | -0.196 (0.352) | -0.080 (0.485)
  Ipsilateral caudate small: Month 18: number analyzed (Participants) | 123 | 109 | 114
  Ipsilateral caudate small: Month 18 | -0.312 (0.383) | -0.273 (0.390) | -0.210 (0.439)
  Ipsilateral putamen small: Month 12: number analyzed (Participants) | 114 | 114 | 95
  Ipsilateral putamen small: Month 12 | -0.178 (0.260) | -0.125 (0.255) | -0.106 (0.219)
  Ipsilateral putamen small: Month 18: number analyzed (Participants) | 123 | 109 | 114
  Ipsilateral putamen small: Month 18 | -0.208 (0.252) | -0.150 (0.260) | -0.179 (0.270)
  Contralateral caudate small: Month 12: number analyzed (Participants) | 114 | 114 | 95
  Contralateral caudate small: Month 12 | -0.256 (0.328) | -0.183 (0.332) | -0.145 (0.363)
  Contralateral caudate small: Month 18: number analyzed (Participants) | 123 | 109 | 114
  Contralateral caudate small: Month 18 | -0.291 (0.330) | -0.263 (0.370) | -0.248 (0.398)
  Contralateral putamen small: Month 12: number analyzed (Participants) | 114 | 114 | 95
  Contralateral putamen small: Month 12 | -0.066 (0.190) | -0.094 (0.223) | -0.053 (0.304)
  Contralateral putamen small: Month 18: number analyzed (Participants) | 123 | 109 | 114
  Contralateral putamen small: Month 18 | -0.115 (0.190) | -0.076 (0.197) | -0.128 (0.209)

19. Secondary Outcome: Time to Start of Symptomatic Treatment (ST)
Description: Time to start of symptomatic treatment (ST) within the 18-month period.
Time Frame: Baseline to Month 18
Population: as for outcome 15
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 163 | 164 | 164
months | 10.58 [9.6242 to 11.5456] | 11.59 [10.6084 to 12.5623] | 11.80 [10.8312 to 12.7735]
Statistical Analysis 1: Comparison: Placebo vs UCB0599 180 mg/Day; Test type: Superiority; p = 0.124, Wald Chi-square; Difference in RMET = 1.00, 95% CI 2-sided [-0.27 to 2.27] — Results were obtained from a generalized linear model for the RMET, with gender and age at baseline as covariates and treatment group as the effect of interest
Statistical Analysis 2: Comparison: Placebo vs UCB0599 360 mg/Day; Test type: Superiority; p = 0.064, Wald Chi-sqaure; Difference in RMET = 1.22, 95% CI [-0.07 to 2.51] — [estimate comment as in outcome 19, analysis 1]

20. Secondary Outcome: Symptomatic Treatment (ST) Intake
Description: Cumulative number of participants on symptomatic treatment (ST) at 18 months are reported.
Time Frame: Month 18
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 153 | 139 | 140
Participants | 111 | 89 | 88

21. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. A TEAE is defined as any AE with a start date on or after the first dose of treatment or any unresolved event already present before administration of treatment that worsens in intensity following exposure to the treatment.
Time Frame: From Baseline up to 30 days of safety follow-up after the last dose of the study drug (up to 19 months)
Population: Safety set included all randomized study participants who receive at least a partial dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 164 | 165 | 164
percentage of participants | 87.8 | 86.7 | 87.2

22. Secondary Outcome: Percentage of Participants With Serious TEAEs
Description: Serious adverse event: Death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: From Baseline up to 30 days of safety follow-up after the last dose of the study drug (up to 19 months)
Population: Safety set included all randomized study participants who receive at least a partial dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 164 | 165 | 164
percentage of participants | 5.5 | 7.9 | 8.5

23. Secondary Outcome: Percentage of Participants With TEAEs Leading to Participant Withdrawal
Description: as for outcome 21
Time Frame: From Baseline up to 30 days of safety follow-up after the last dose of the study drug (up to 19 months)
Population: Safety set included all randomized study participants who receive at least a partial dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
Number analyzed (Participants) | 164 | 165 | 164
percentage of participants | 2.4 | 10.9 | 9.8

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days of safety follow-up after the last dose of the study drug (up to 19 months)
Description: Safety analysis set included all randomized study participants who received at least a partial dose of study medication.
Arm/Group | Placebo | UCB0599 180 mg/Day | UCB0599 360 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/164 | 1/165 | 1/164
Serious Adverse Events (participants affected / at risk) | 9/164 | 13/165 | 14/164
Other Adverse Events (participants affected / at risk) | 102/164 | 97/165 | 89/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=164) | UCB0599 180 mg/Day (N=165) | UCB0599 360 mg/Day (N=164)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=164) | UCB0599 180 mg/Day (N=165) | UCB0599 360 mg/Day (N=164)
Nausea (Gastrointestinal disorders) | 8 (15) | 12 (14) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 10 (18) | 9 (10)
Constipation (Gastrointestinal disorders) | 14 (14) | 7 (7) | 8 (9)
Fatigue (General disorders) | 12 (14) | 13 (15) | 7 (7)
COVID-19 (Infections and infestations) | 35 (38) | 22 (23) | 32 (33)
Urinary tract infection (Infections and infestations) | 15 (20) | 18 (26) | 12 (14)
Nasopharyngitis (Infections and infestations) | 19 (20) | 14 (16) | 14 (15)
Influenza (Infections and infestations) | 10 (10) | 6 (7) | 14 (15)
Fall (Injury, poisoning and procedural complications) | 9 (9) | 17 (22) | 12 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 15 (19) | 12 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (22) | 14 (14) | 4 (4)
Headache (Nervous system disorders) | 16 (17) | 11 (25) | 16 (24)
Rash (Skin and subcutaneous tissue disorders) | 9 (10) | 5 (5) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04658186/Prot_002.pdf
  • Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04658186/SAP_003.pdf